CLINICAL TRIAL: NCT00290134
Title: Preliminary Efficacy and Safety of Fispemifene in the Treatment of Hypogonadism: A 4 Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing Daily Oral Doses of 100, 200, and 300 mg Fispemifene and Placebo
Brief Title: A Preliminary Clinical Study to Evaluate Fispemifene in the Treatment of Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QuatRx Pharmaceuticals Company (Industry)
Collaborators: Hormos Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101-50204
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone
MeSH Terms: conditions — Hypogonadism

INTERVENTIONS:
Drug: Fispemifene once daily for 4 weeks

SUMMARY:
The purpose of this study is to determine whether one or more fispemifene dose regimens are more effective than placebo in the treatment of hypogonadism in older men.

ELIGIBILITY:
Inclusion Criteria:

* Total testosterone level <240 ng/dL
* Serum LH and FSH levels within normal limits

Exclusion Criteria:

* Elevated prolactin
* Evidence of Benign Prostatic Hypertrophy
* History of or current breast cancer, prostate cancer, abnormal DRE or elevated PSA or any other malignancy
* Clinically significant endocrine/metabolic or cardiovascular disease
* Significant polycythemia

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in morning total testosterone levels from baseline to Week 4 (end of therapy)

SECONDARY OUTCOMES:
Change in total testosterone levels from baseline to Weeks 2 and 6
Change in free testosterone, calculated free testosterone, and DHT from baseline to Weeks 2, 4, and 6
Change in SHBG, E2, LH, FSH and inhibin B from baseline to Weeks 2, 4, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Janne Komi, MD, PhD, Study Director — Hormos Medical
Locations (16):
- United States (16):
  - Clinical Research Site, Huntsville, Alabama
  - Clinical Research Site, Modesto, California
  - Clinical Research Site, Aurora, Colorado
  - Clinical Research Site, Waterbury, Connecticut
  - Clinical Research Site, New Port Richey, Florida
  - Clinical Research Site, Tallahassee, Florida
  - Clinical Research Site, Peoria, Illinois
  - Clinical Research Site, Greenbelt, Maryland
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Garden City, New York
  - Clinical Research Site, Poughkeepsie, New York
  - Clinical Research Site, Williamsville, New York
  - Clinical Research Site, Bethany, Oklahoma
  - Clinical Research Site, Greer, South Carolina
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Seattle, Washington

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Assessing the Need for Clinical Trials of Testosterone Replacement Therapy; Liverman CT, Blazer DG, editors. Testosterone and Aging: Clinical Research Directions. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216173/ PMID 25009850
- [Background] Harman SM, Metter EJ, Tobin JD, Pearson J, Blackman MR; Baltimore Longitudinal Study of Aging. Longitudinal effects of aging on serum total and free testosterone levels in healthy men. Baltimore Longitudinal Study of Aging. J Clin Endocrinol Metab. 2001 Feb;86(2):724-31. doi: 10.1210/jcem.86.2.7219. PMID 11158037
- [Background] Feldman HA, Longcope C, Derby CA, Johannes CB, Araujo AB, Coviello AD, Bremner WJ, McKinlay JB. Age trends in the level of serum testosterone and other hormones in middle-aged men: longitudinal results from the Massachusetts male aging study. J Clin Endocrinol Metab. 2002 Feb;87(2):589-98. doi: 10.1210/jcem.87.2.8201. PMID 11836290
- [Background] Nieschlag E, Swerdloff R, Behre HM, Gooren LJ, Kaufman JM, Legros JJ, Lunenfeld B, Morley JE, Schulman C, Wang C, Weidner W, Wu FC; International Society of Andrology (ISA); International Society for the Study of the Aging Male (ISSAM); European Association of Urology (EAU). Investigation, treatment and monitoring of late-onset hypogonadism in males. ISA, ISSAM, and EAU recommendations. Eur Urol. 2005 Jul;48(1):1-4. doi: 10.1016/j.eururo.2005.04.027. No abstract available. PMID 15951102
- [Background] Morales A, Lunenfeld B; International Society for the Study of the Aging Male. Investigation, treatment and monitoring of late-onset hypogonadism in males. Official recommendations of ISSAM. International Society for the Study of the Aging Male. Aging Male. 2002 Jun;5(2):74-86. No abstract available. PMID 12198738